CLINICAL TRIAL: NCT05627271
Title: Understanding the 'Wearing Off' Effect From Disease-modifying Therapies (DMT) in Patients With Multiple Sclerosis: an Interview Based Study Among Patients and Clinicians
Brief Title: The 'Wearing Off' Effect of DMT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G2012
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; ocrelizumab; Ocrevus; natalizumab; Tysabri; ofatumumab; Kesimpta; NIS
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab; Natalizumab; ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- ocrelizumab: patients prescribed with ocrelizumab
  Interventions: Other: ocrelizumab
- natalizumab: Patients prescribed with natalizumab
  Interventions: Other: natalizumab
- ofatumumab: Patients prescribed with ofatumumab
  Interventions: Other: ofatumumab

INTERVENTIONS:
Other: ocrelizumab — Non-interventional, cross-sectional, qualitative study. There is no treatment allocation. Patients prescribed with Disease-modifying therapy in the commercial setting are eligible to enroll into this study.
  Other Names: Ocrevus
  Groups: ocrelizumab
Other: natalizumab — Non-interventional, cross-sectional, qualitative study. There is no treatment allocation. Patients prescribed with Disease-modifying therapy in the commercial setting are eligible to enroll into this study.
  Other Names: Tysabri
  Groups: natalizumab
Other: ofatumumab — Non-interventional, cross-sectional, qualitative study. There is no treatment allocation. Patients prescribed with Disease-modifying therapy in the commercial setting are eligible to enroll into this study.
  Other Names: Kesimpta
  Groups: ofatumumab

SUMMARY:
This is a non-interventional, cross-sectional, qualitative study in which patients diagnosed with MS and clinicians with experience treating MS will be interviewed regarding patient experiences with the wearing off effect from ocrelizumab, natalizumab, and ofatumumab

ELIGIBILITY:
Inclusion Criteria:

Patients who attend the following criteria will be included:

1. Age ≥18;
2. Current resident of the country of interest (i.e., Germany, the UK, or the US);
3. Relapsing-remitting MS diagnosis confirmed by a clinician;
4. Currently taking at least one of the following DMTs for MS after the maintenance phase: ocrelizumab (Ocrevus®), natalizumab (Tysabri®), or ofatumumab (Kesimpta®);
5. Two or more consecutive ocrelizumab doses (Six or more consecutive natalizumab doses or Six or more consecutive ofatumumab doses);
6. Follow the approved dosing regimen (Ocrelizumab: every six months or Natalizumab: every month or Ofatumumab: every month);
7. Experienced reoccurring symptoms towards the end of the dosing cycle (i.e., the wearing off effect);
8. Willing and able to provide informed consent via a weblink, indicating they understand the study purpose and procedures and are willing to participate;
9. Able to read, understand, and communicate in English or German;
10. Willing and able to participate in a phone/web-based (remote) one-on-one interview, and to be audio-recorded;
11. Have an e-mail address and will have access to a computer or smartphone at the time of the interview to complete the electronic consent form.

Clinicians who attend the following criteria will be included:

1. Currently practices in one of the target countries (i.e., Germany, the UK, or the US);
2. Is a licensed clinician with a specialty in neurology;
3. Has prescribed at least one of the following DMTs within the last year: ocrelizumab (Ocrevus®), natalizumab (Tysabri®), or ofatumumab (Kesimpta®);
4. Has treated at least 16 MS patients within the last month;
5. Is personally responsible for treatment decisions for their patients;
6. Has followed patients treating MS with any of the three DMTs for a. Two or more consecutive ocrelizumab doses or b. Six or more consecutive natalizumab doses. c. Six or more consecutive ofatumumab doses;
7. Has treated patients who have experienced specific reoccurring symptoms towards the end of the dosing cycle (i.e., the wearing off effect);
8. Willing and able to provide informed consent via a weblink, indicating they understand the study purpose and procedures and are willing to participate;
9. Willing and able to participate in a phone/web-based interview, and to be audio-recorded.
10. Able to read, understand, and communicate in English

Exclusion Criteria:

Patients will be excluded from the enrollment if:

1. Has a diagnosis of clinically isolated MS syndrome, primary progressive MS, or secondary progressive MS;
2. Currently participates in an interventional MS clinical trial.

Clinicians will be excluded from the enrollment if are currently involved as a key opinion leader or receives funding from one of the drug manufacturers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with MS and clinicians with experience treating MS from Germany, UK, and US
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with key symptoms associated with the wearing off effect | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Number of participants with the following recurring symptoms will be collected:
  * Fatigue
  * Physical Pain
  * Mobility issues or walking difficulties
  * Numbness or sensory issues
  * Cognitive difficulties
  * Weakness
  * Spasms
  * Balance disturbance or dizziness
  * Blurry vision or visual impairment
  * Others

SECONDARY OUTCOMES:
Severity of wearing off effect symptoms | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Based on qualitative score rating
Detailed language used to describe the experience of wearing off effect | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Terms used to describe times when patients MS "gets better" and when it "gets worse" will be collected.
Number of participants switching from one therapy to another due to wearing off effect | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Number of participants switching from one therapy to another due to wearing off effect will be collected
Number of participants who changed the dosing/infusion schedules due to wearing off effect | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Number of participants who changed the dosing/infusion schedules due to wearing off effect will be collected
Dissimilarities of clinician' and patients' views of wearing off effect | Assessed at the time of interview with lookback period from time of first MS diagnosis, up to 3 months
  Assessed qualitatively via concept coding techniques

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No